CLINICAL TRIAL: NCT06365021
Title: Acceptance and Commitment Therapy for Individuals With Syndromic and Subsyndromic Depression in Bipolar Mood Disorder: A Controlled and Randomized Clinical Trial
Brief Title: ACT for Syndromic and Subsyndromic Depression in Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beny Lafer (Other)
Responsible Party: Sponsor-Investigator, Beny Lafer, Principal Investigator, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88887.687583/2022-00
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder
Keywords: Acceptance and Commitment Therapy; Bipolar Disorder; Psychotherapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Participants in the clinical group will receive usual pharmacological treatment and undergo a protocol of 12 Acceptance and Commitment Therapy sessions, in group format, during 3 months. The intervention will be held weekly, with an estimated duration of 2 hours for each session, in addition to the participants' regular drug treatment. Scales are administered at the beginning and end of treatment, with follow-ups after 6, 9 and 12 months.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Psychoeducation (Experimental): Participants in the control group will usual pharmacological treatment and 3 sessions of Psychoeducation, in group format. Scales are administered at the beginning and end of treatment, with follow-ups after 6, 9 and 12 months.
  Interventions: Other: Bipolar Disorder Psychoeducation Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The ACT protocol for this study was developed by ACT psychologist Tatiana Cohab Khafif specifically for this study and for Bipolar Patients. It is a 12-session protocol that combines psychoeducation elements, mindfulness exercises, experiential exercises, discussions and group processes, homework assignments, and flexible repertoire modeling and training. The protocol is designed to fit into a single trimester. It covers all the basic aspects of Bipolar Disorder and the six processes of ACT.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy
Other: Bipolar Disorder Psychoeducation Therapy — The psychoeducation protocol for this study was developed by clinical psychologist Tatiana Cohab Khafif specifically for this study and for Bipolar Patients. It is a 3-session protocol that combines psychoeducation elements, mindfulness exercises, and discussions regarding the main aspects and symptoms of BD. The protocol is designed to fit into a single month, and has a specifically brief format in order for it not to crossover with psychotherapy. It covers all the basic aspects of Bipolar Disorder.
  Arms: Psychoeducation

SUMMARY:
The goal of this clinical trial is to test the efficacy of Acceptance and Commitment Therapy (ACT) as a psychotherapeutic treatment for patients with Bipolar Disorder (BD). The following questions will be investigated:

* The efficacy of ACT in reducing depressive symptoms in patients with BD.
* The efficacy of ACT in improving the quality of life in patients with BD.
* The efficacy of ACT in improving functionality in patients with BD.
* The efficacy of ACT in improving sleep quality in patients with BD.
* The efficacy of ACT in improving psychological flexibility in patients with BD

Participants in the clinical group will undergo 12, 2 hours, weekly sessions of Acceptance and Commitment Therapy, in addition to their regular pharmacological treatment.

Participants in the control group will undergo 3, 2 hours, weekly sessions of Bipolar Disorder Psychoeducation Therapy, in addition to their regular pharmacological treatment.

Scales and assessments will be used to measure study outcomes on 5 different time-points: pre-intervention (month 0), post-intervention (month 3), follow-up 1 (month 6), follow-up 2 (month 9), follow-up 3 (month 12). Mood scales will be assessed every 2 weeks for the duration of treatment and every 4 weeks during the additional 12 week follow-up period.

Results will be compared among both groups to assess the effectiveness of Acceptance and Commitment Therapy as an intervention for syndromic and sub-syndromic depression in bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a serious psychiatric disorder characterized by recurrent episodes of mania and depression. The treatment of BD includes a combination of pharmacological medications and psychotherapy to manage episodes and prevent recurrence.

Acceptance and Commitment Therapy (ACT) is an evidence-based psychotherapy. Although there is ample evidence for the efficacy of ACT in the treatment of psychiatric disorders, the literature on ACT for BD is still scarce.There are only five published studies, with three of them being pilot studies.

The present study is justified by the importance to fill a gap in the literature, by aiming to evaluate the effectiveness of ACT as a psychotherapeutic intervention for BD patients and to understand its possible effects mood, quality of life, functionality, sleep, and psychological flexibility on this population.

Main Objective:

To investigate the effectiveness of ACT, in improving syndromic and sub-syndromic depressive symptoms in patients with BD.

Specific objectives:

1. To investigate the efficacy of ACT for improving the quality of life in patients with BD.
2. To investigate the efficacy of ACT in improving functionality in patients with BD.
3. To investigate the efficacy of ACT in improving sleep quality in patients with BD.
4. To investigate the efficacy of ACT in improving psychological flexibility in patients with BD.

Material and Methods:

All participants will be recruited from patients regularly enrolled at the Bipolar Disorder Program - PROMAN - outpatient clinic at Hospital das Clínicas, Faculdade de Medicina, Universidade de São Paulo. Participants will have access to the Informed Consent Form (ICF), and only those who agree to participate will be included in the study. Randomization Individuals with Bipolar Disorder recruited for the research will be randomized to the ACT arm or Usual Treatment arm through the Online Randomization software.

Procedures:

1. Recruitment will take place in the outpatient clinic of the Bipolar Disorder Program (PROMAN) of the HC-FMUSP Psychiatric Institute and online through the Hospital's social medias.
2. Interested individuals will undergo an initial screening to verify eligibility based on the selection criteria established in the study.
3. Individuals who meet the inclusion criteria will undergo a psychiatric evaluation based on the Standardized Structured Clinical Diagnostic Interview for DSM IV - Axis I Disorders (M.I.N.I.). and complete the initial phase (pre-treatment) instruments via the REDCap platform.
4. Included participants will be randomized into ACT or Psychoeducation group.
5. Participants will be contacted by email or text message with informations regarding the start of treatment.
6. Throughout the intervention, Mood scales (YMRS and MADRS) will be administered periodically (every two weeks)
7. At the end of the intervention, the same assessments administered at baseline will be repeated, as well as at 6, 9 and 12-month follow-ups.

For control purposes, medication changes will be monitored using the MRTF Scale, which allows monitoring of the frequency, type, and reasons for changes in dosages and medications during the intervention protocol. Throughout the study, participants in both groups will continue to receive their usual pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder type I and II according to DSM V
* Presence of depressive symptoms (MADRS>12)
* Not undergoing psychotherapy
* Availability to attend in-person group therapy sessions
* Signing consent form

Exclusion Criteria:

* Organic mental disorder
* Presence of manic or hypomanic symptoms (YMRS>12)
* Currently undergoing psychotherapy (not able to pause during the study)
* Major medication change in last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Scale | Baseline, during treatment every 2 weeks, post-treatment (week 12), in between assessments every 4 weeks, and follow-ups (6, 9 and 12 months)
  Minimum value: 0 (better) Maximum value: 60 (worse)
Young Mania Rating Scale | Baseline, during treatment every 2 weeks, post-treatment (week 12), in between assessments every 4 weeks, and follow-ups (6, 9 and 12 months)
  Minimum value: 0 (better) Maximum value: 54 (worse)

SECONDARY OUTCOMES:
Functional Assessment Staging Tool | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum value: 0 (better) Maximum value: 72 (worse)
World Health Organization Quality of Life Brief Scale | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum value: 0 (worse) Maximum value: 100 (better)
Pittsburgh Sleep Quality Index | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum Value: 0 (better) Maximum Score: 21 (worse)
Psychological Flexibility Questionnaire | Baseline, during treatment weekly, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum value: 7 (worse) Maximum value: 49 (better) Higher scores mean a better outcome

OTHER OUTCOMES:
Generalized Anxiety Disorder 7-item Scale | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum value: 0 (better) Maximum value: 21 (worse)
Medication Recommendation Tracking Form | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Tracks patient medication use and dosage. There is no score.
Regulatory Satisfaction Alertness Timing Efficiency Duration | Baseline, post-treatment (week 12), and follow-ups (6, 9 and 12 months)
  Minimum Value: 0 (worse) Maximum Value: 18 (better)

CONTACTS AND LOCATIONS:
Overall Officials: Beny Lafer, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Tatiana Cohab Khafif, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided